CLINICAL TRIAL: NCT06816147
Title: Empowering Healthy Lifestyle Behavior Through Personalized Intervention Portfolios to Prevent and Control Obesity in the Elderly
Brief Title: HealthyW8_60+ Pilot
Acronym: HealthyW8
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Luxembourg Institute of Health (Other Government)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 101080645
Record Dates: First submitted 2024-12-05; First posted 2025-02-10 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-09

CONDITIONS: Obesity Prevention
Keywords: Obesity; BMI; overweight; life style recommender solution
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Intervention Model Description: The project is a pilot study. It is a single-group study where participants will be their own control (i.e. outcome measures at the end of study will be compared to baseline). 30 participants will be included. It consists of samples and data collection, together with a mobile application that allows dispensing an intervention that will last 3 months.
  This pilot study will be longitudinal design without a control group. A later trial that is planned for the following year will focus further on biological endpoints and will be randomized. In this present pilot study, investigators aim to assess mainly the user-friendliness of the HLRS, and gather first evidence that the intervention can indeed produce healthier lifestyle patterns. Should the participants complete the study, the individual duration will be 3 months. Investigators foresee that, in total, given the various enrolments of the participants, up to 6 months may be necessary for all participants to complete the entire study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participant from the general population living in Luxembourg free of manifest diagnosed diseases (Experimental): The following clinical visits and data collection points will be set up within the study:
  1. Enrollment visit: the participant will sign the informed consent, the eligibility of the participant will be evaluated based on anthropometric measures, a urine spot sample, as well as general questionnaire. If found eligible, the participant can continue the study
  2. Baseline visit: a number of questionnaires will be filled out by the participant, anthropometric data will be obtained, and a urine and blood sample will be taken, and a stool sample will be provided
  3. Intermediate follow-up: this will consist of a phone interview or physical meeting
  4. Final visit: a number of questionnaires will be filled anthropometric data, urine, blood and stool will be collected
  Interventions: Other: Investigators will evaluate the acceptance and adherence to a healthy lifestyle recommender solution (HLRS), a digital app, among participants

INTERVENTIONS:
Other: Investigators will evaluate the acceptance and adherence to a healthy lifestyle recommender solution (HLRS), a digital app, among participants — The intervention will include collecting blood, stool, urinary samples as well as measuring anthropometrics and collecting data (socio-demographics, general health, well-being, PA, and eating patterns, among others) via questionnaires completed in part from a mobile application.

SUMMARY:
This pilot study will focus on men and women aged ≥60 years for a period of 3 months during which each participant will use the HLRS. The primary purpose is to study whether the HLRS, reflecting a multi-component intervention, is well accepted by the participant, has a decent adherence (i.e., user time of the app). In addition, investigators will study the feasibility of the design, i.e. whether the overall design is well suited to the participants, in order to improve their lifestyle, e.g., dietary habits and PA, among others. Secondary outcomes related to the feasibility approach include dietary habits, PA patterns, and selected plasma and urinary endpoints. This pilot study will be of longitudinal design without a control group. A later trial that is planned for the following year will focus further on biological endpoints and will be randomized. In this present pilot study, investigators aim to assess mainly the user-friendliness of the HLRS, and gather first evidence that the intervention can indeed produce healthier lifestyle patterns.

The study's primary objective is to determine whether the developed HLRS can be successfully applied to the target population (men and women aged ≥60 years) and whether they use it frequently during the study and are satisfied with the HLRS.

Secondly, investigators will study whether the assessment of endpoints required for the later and separately planned ensuing long-term study can be well assessed within the study and if, despite the limited time of the intervention duration, the intervention will be able to preliminary improve specific markers related to the risk of obesity and associated comorbidities. This will entail anthropometric measures to assess changes in body mass and body fat in addition to the primary and secondary objectives.

DETAILED DESCRIPTION:
The number of people struggling with overweight and obesity continues to grow in most countries worldwide, despite varied measures trying to limit the further progress of this pandemic. In Luxembourg, at present, about 26% of the adult population is considered as having obesity(BMI>30 kg/m²), and the associated health costs have been estimated at 1.4% of the GDP or about 930 Mio. USD for Luxembourg. Similar numbers are prevalent in other European countries.

The ongoing problem of high obesity rates has resulted in the creation of a pan-European project HealthyW8 (www.healthyw8.eu), funded by the European Union and in which the Luxembourg Institute of Health (LIH) is the coordinator.

The study described in this application is therefore motivated by the project's main objectives, which entails, among other, a total of 22 pilot trials in various European countries to be conducted. This application concerns only the activities planned in Luxembourg.

With the HealthyW8_65+ Pilot project, investigators have focused on population groups at risk of developing obesity, due to undergoing transitions in their lifestyle. Among the populations at risk are older adults as, categorized as having an age of equal to or above 65 years. As emphasized in the literature, older adults constitute a growing fraction of our society, with likely high associated healthcare costs, whose change to a more sedentary lifestyle upon retirement adds an additional risk factor, especially for sarcopenic obesity and related comorbidities, i.e., low muscle mass and consequences.

As innovative solutions to combat the trend toward increasing overweight and obesity in our society are much in need, the present study aims to employ the developed healthy lifestyle recommender solution (HLRS), which is at the center of a digital application for mobile phones. This HLRS intends to address various factors known to constitute main risks for developing obesity, including dietary patterns, physical activity (PA), and psychological/behavioral ones, among other lifestyle factors, such as sleep patterns, while also considering socio-demographic aspects. Our approach addresses several of the shortcomings of existing apps by catering to individuals with low interest in healthy lifestyles and try to motivate them via nudges and gamifications and organized information sessions to participate.

The pilot study will primarily focus on usability and user experience of the HLRS. An accurate assessment of food intake will be ensured through validated semi-quantitative FFQs and user feedback from the HLRS regarding meals that have been consumed. It is important to note, however, that there will be a secondary outcome, i.e. to test the operational feasibility of the study. This includes collecting biological samples, their measuring and shipment to partners outside Luxembourg. This is important, as this pilot study will be followed by a long term study, i.e. employing the same developed HLRS, but then targeting rather metabolic changes.

ELIGIBILITY:
Inclusion Criteria:

Individuals aged 60 or older:

* both males/females, general free-living population,
* residing in Luxembourg,
* having normal weight or being overweight, i.e., with a BMI between 18.5 ; 30 kg/m², which is considered a risk factor for developing obesity,
* owning a smartphone.

Exclusion Criteria:

* With known manifest chronic diseases that prohibits participation in the study (e.g., cancer, Parkinson's),
* Persons with cognitive diseases (Alzheimer's) or those who are not able to lead an independent life,
* Persons following a strict diet (on their own or advised by their physician),
* Particular population groups, such as prisoners, the mentally disabled, or groups whose ability to give voluntary informed consent may be in question.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-19 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Health Lifestyle Recommender System adherence time | 3 month intervention period from baseline (Day 1) to final measurement (Day 90)
  Adherence time (daily and weekly usage time in minutes) will be measured by tracking through user log-data, with analysis of any significant changes in usage comparing baseline with final measurement.
Health Lifestyle Recommender system user experience | 3 month intervention period from baseline (Day 1) to final measurement (Day 90)
  User experience corresponds to the points achieved in the User Experience Questionnaire (UEQ+, 26 items). This questionnaire analyses the attractiveness, perspicuity, efficiency, dependability, stimulation and novelty of a new product (in this case HLRS).
  The UEQ contains 26 items. Each item is evaluated with a 7-point Likert scale (-3 to 3 points). Then the product is classified as excellent (3 points) or bad (-3 points).

SECONDARY OUTCOMES:
Anthropometric measurements (1/4) | 3 month intervention period from baseline (Day 1) to final measurement (Day 90)
  Body mass index (kg/m^2) will be calculated with weight (kg) and height (m).
Anthropometric measurements (2/4) | 3 month intervention period from baseline (Day 1) to final measurement (Day 90)
  Waist and hip circumference (cm) measure and thigh circumference (cm) obtained with a tape
Anthropometric measurements (3/4) | 3 month intervention period from baseline (Day 1) to final measurement (Day 90)
  Body fat percentage determined by a bioelectrical impedance scale (Tanita)
Anthropometric measurements (4/4) | 3 month intervention period from baseline (Day 1) to final measurement (Day 90)
  Visceral body fat (cm2) determined by anthropometric measurements including weight, height, waist circumference and thigh circumference (https://www.lih.lu/en/visceral-fat-calculator/).
Physical activity and fitness (1/4) | 3 month intervention period from baseline (Day 1) to final measurement (Day 90)
  24-hour movement obtained by accelerometer to calculate metabolic equivalent of task (METs)
Physical activity and fitness (2/4) | 3 month intervention period from baseline (Day 1) to final measurement (Day 90)
  International Physical Activity Questionnaire to obtain METS and minutes per week of physical activity. The higher the METs the higher the physical activity intensity.
Physical activity and fitness (3/4) | 3 month intervention period from baseline (Day 1) to final measurement (Day 90)
  Hand-grip strength (kg) to assess the cardio-physiological fitness.
Physical activity and fitness (4/4) | 3 month intervention period from baseline (Day 1) to final measurement (Day 90)
  Quick step-up test (number of step-ups achieved) to assess the cardio-physiological fitness.
Clinical measurements | 3 month intervention period from baseline (Day 1) to final measurement (Day 90)
  Blood pressure is going to be measure with a baumanometer. During the measurement it is obtained two number, the first number is the systolic pressure (mmHg) and the second one is the diastolic pressure (mmHg)
Biochemical analysis (1/12) | 3 month intervention period from baseline (Day 1) to final measurement (Day 90)
  Biochemical analysis such as the lipid profile including total-cholesterol, LDL-C, HDL-C, and triglycerides (mg/dL); glucose metabolism including fasting blood glucose (mg/dL); vitamin E (mg/dL), CRP (mg/dL), hemoglobin (mg/dL)
Biochemical analysis (2/12) | 3 month intervention period from baseline (Day 1) to final measurement (Day 90)
  It will be analyzed nutrition related parameters such as albumin (g/dL) and prealbumin (g/dL)
Biochemical analysis (3/12) | 3 month intervention period from baseline (Day 1) to final measurement (Day 90)
  Hormones including ghrelin (pg/mL) and inflammation biomarkers such as IL-6 (pg/mL) and TNF-α (pg/mL) will be analyzed
Biochemical analysis (4/12) | 3 month intervention period from baseline (Day 1) to final measurement (Day 90)
  Glucose metabolism will be analysed by glycated haemoglobin (HbA1c, %)
Biochemical analysis (5/12) | 3 month intervention period from baseline (Day 1) to final measurement (Day 90)
  Insulin resistance will be analysed with Homeostatic Model Assessment for Insulin Resistance) HOMA-IR (no units)
Biochemical analysis (6/12) | 3 month intervention period from baseline (Day 1) to final measurement (Day 90)
  Total carotenoids (µmol/L)
Biochemical analysis (7/12) | 3 month intervention period from baseline (Day 1) to final measurement (Day 90)
  Hormones such as leptin (ng/mL) and oxidative stress biomarkers like F2-isoprostanes (ng/mL)
Biochemical analysis (8/12) | 3 month intervention period from baseline (Day 1) to final measurement (Day 90)
  Adiponectin (µg/mL)
Biochemical analysis (9/12) | 3 month intervention period from baseline (Day 1) to final measurement (Day 90)
  Malondialdehyde (nmol/L)
Biochemical analysis (10/12) | 3 month intervention period from baseline (Day 1) to final measurement (Day 90)
  DNA/RNA breakdown products (µg/L)
Biochemical analysis (11/12) | 3 month intervention period from baseline (Day 1) to final measurement (Day 90)
  Antioxidant capacity FRAP (µmol/L)
Biochemical analysis (12/12) | 3 month intervention period from baseline (Day 1) to final measurement (Day 90)
  ABTS (mg/L)
Diet analysis (1/3) | 3 month intervention period from baseline (Day 1) to final measurement (Day 90)
  The healthiness of the diet will be assessed using the Healthy Eating Index (HEI). The HEI employs a scoring system to evaluate a set of foods, with scores ranging from 0 to 100. An ideal overall HEI score of 100 indicates that the set of foods aligns with key dietary recommendations and dietary patterns.
Diet analysis (2/3) | 3 month intervention period from baseline (Day 1) to final measurement (Day 90)
  Food frequency questionnaire (FFQ) comprises 151 items designed to gather information on food intake frequencies including daily, weekly and monthly consumption. The 24-hour recall method obtains the intake from the past 24 hours. After analyzing the data, the total kilocalories and grams of carbohydrates, protein and lipids consumed during that specific period are determined.
Diet analysis (3/3) | 3 month intervention period from baseline (Day 1) to final measurement (Day 90)
  Chrononutrition questionnaire will be administered to determine the times of the day participants consume their meals and frequency (days per week) in which they eat breakfast, lunch, dinner and snacks. This tool provides a qualitative analysis of dietary habits. Therefore, it does not provide a numerical score or points.
Lifestyle measurements(1/9) | 3 month intervention period from baseline (Day 1) to final measurement (Day 90)
  Depression will be assessed using the Patient Health Questionnaire-9 (PHQ-9), a validated tool measuring the severity of depression. The PHQ-9 consists of 9 items, each scored on a scale from 0 to 3, based on the frequency of symptoms experienced over the past two weeks. The total score ranges from 0 to 27, with higher scores indicating greater severity of depression. A score between 20 and 27 suggests severe depression.
Lifestyle measurements (2/9) | 3 month intervention period from baseline (Day 1) to final measurement (Day 90)
  Mood and emotion will be assessed using the Positive and Negative Affect Schedule (PANAS). This instrument consists of 20 items, divided into two subscales: Positive Affect (PA) and Negative Affect (NA). Each item is rated on a 5-point Likert scale, ranging from 1 (very slightly or not at all) to 5 (extremely). To calculate the scores, sum the ratings for the items in each subscale separately. Higher scores indicate greater levels of the corresponding affect. For example, a higher PA score reflects higher levels of positive affect, while a higher NA score indicates higher levels of negative affect.
Lifestyle measurements (3/9) | 3 month intervention period from baseline (Day 1) to final measurement (Day 90)
  Psychological hardiness, encompassing aspects of commitment, control, and challenge, will be assessed using the Dispositional Resilience Scale (DRS-15). This 15-item self-report instrument measures an individual's resilience and ability to cope with stress. Each item is rated on a 4-point Likert scale, ranging from 0 ("not at all true") to 3 ("completely true"). The DRS-15 provides a total hardiness score, with higher scores indicating greater psychological hardiness.
Lifestyle measurements (4/9) | 3 month intervention period from baseline (Day 1) to final measurement (Day 90)
  Sleep disturbances will be assessed using the Pittsburgh Sleep Quality Index (PSQI). This instrument consists of 19 self-rated questions. Each component is scored on a scale from 0 to 3, with higher scores indicating more severe sleep disturbances. The component scores are then summed to produce a global score ranging from 0 to 21; higher global scores denote poorer sleep quality.
Lifestyle measurements (5/9) | 3 month intervention period from baseline (Day 1) to final measurement (Day 90)
  Mediterranean eating patterns will be assessed by administrating the Mediterranean Diet Adherence Screener (MEDAS-14). This is a 14 item questionnaire of food consumptions to evaluate the amount of 12 main components consumed and two food habits related to the MD. Each of the 14 item is scored with 1 point or 0 points (total score of 14 points), depending on whether participants are adherent to each of the MD (1 point) or not (0 points). The higher the score the higher the adherence to the Mediterranean diet.
Lifestyle measurements (6/9) | 3 month intervention period from baseline (Day 1) to final measurement (Day 90)
  To evaluate participants' subjective experiences related to a specific activity, the Intrinsic Motivation Inventory (IMI) will be administered. The IMI comprises multiple sections, each containing various statements. Participants will respond to each statement using a 5-point Likert scale. To score the IMI, calculate the subscale scores by averaging the item scores within each subscale. A higher score indicates a greater presence of the concept described by the subscale name. For instance, a higher score on the Pressure/Tension subscale suggests that the individual felt more pressured and tense.
Lifestyle measurements (6/9) | 3 month intervention period from baseline (Day 1) to final measurement (Day 90)
  Smoking behavior will be assessed using the Fagerström Test for Nicotine Dependence. This instrument consists of six questions designed to evaluate the intensity of physical addiction to nicotine. Each question is scored on a scale from 0 to 1 or 0 to 3, depending on the response options. The total score is calculated by summing the individual item scores, resulting in a range from 0 to 10. Lower total scores indicate less nicotine dependence, while higher scores reflect greater dependence.
Lifestyle measurements (7/9) | 3 month intervention period from baseline (Day 1) to final measurement (Day 90)
  Alcohol consumption, drinking behaviors, and alcohol-related problems will be assessed by administrating the Alcohol Use Disorders Identification Test (AUDIT). This instrument is a 10-item screening tool. The range of possible scores is from 0 to 40 where 0 indicates an abstainer who has never had any problems from alcohol.
Lifestyle measurements (9/9) | 3 month intervention period from baseline (Day 1) to final measurement (Day 90)
  Personal traits will be assessed by administrating the Big Five Inventory (BFI) with 10 items. The BFI-10 is a scale measuring the Big Five personality traits Extraversion, Agreeableness, Conscientiousness, Emotional Stability, and Openness. To score the BFI-10, sum the responses for each trait, ensuring that reverse-scored items are appropriately adjusted. Higher scores indicate a greater association with that particular trait.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical and Epidemiological Investigation Center CIEC- LCTR, Luxembourg, Luxembourg